CLINICAL TRIAL: NCT05219227
Title: Effect of 12 Session of Laser Acupuncture Augmented by Abdominal Exercises on Abdominal Fat in Obese Breast-feeding Women
Brief Title: Effect of Laser Acupuncture Augmented by Abdominal Exercises on Abdominal Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Rafat, lecturer of physical therapy, basic science department, faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC
Record Dates: First submitted 2021-12-06; First posted 2022-02-02 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Obesity, Abdominal
Keywords: obesity; laser acupuncture; abdominal exercises
MeSH Terms: conditions — Obesity, Abdominal; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- body fat mass (BFM) (Experimental): body fat mass will be measured before and after interventions
  Interventions: Other: laser acupuncture and abdominal exercises
- Body mass index (BMI) (Experimental): BMI will be calculated before and after interventions
  Interventions: Other: laser acupuncture and abdominal exercises

INTERVENTIONS:
Other: laser acupuncture and abdominal exercises — laser acupuncture on certain point on the abdomen The following abdominal acupuncture points were irradiated: Cv 8 (Shenque), St 25 (Tianshu, bilateral), and Sp 15 (Daheng
  , bilateral). The laser irradiations were applied directly to the skin of the points with a perpendicular beam. 478 J/cm2
  Abdominal exercises:
  Types of abdominal exercises:
  1. Static abdominal exercises:
  2. Dynamic abdominal exercises:
     * Hip shrugging exercise from crook lying position:
     * Lateral flexion of the trunk from crook lying position:
     * Antero-posterior flexion of the trunk from crook lying position:

SUMMARY:
the aim of study is to investigate the effect of laser acupuncture and abdominal exercises on abdominal fat in breast feeding women

DETAILED DESCRIPTION:
Forty breast feeding women aged between 20 and 35 years will recruited to the study in the women health department faculty of physical therapy clinic, kafr el sheikh university , Egypt. The evaluation procedures will explained to each participant. participants will be divided into two groups Group A : received laser acupuncture, diet modification and abdominal exercises Group B: received diet modification and abdominal exercises only

Out come measurement BW, BMI, body fat mass (BFM), body fat percent, waist girth, hip girth, and waist-to-hip ratio (WHR) were measured at baseline and the end of treatment. BW, BMI, BFM, and body fat percent were measured using the body composition analyzer (Model Inbody 3.0, Republic of Korea).

ELIGIBILITY:
Inclusion Criteria:

* All participants are free from any medical problems such as diabetes mellitus, hypertension and thyroid dysfunction.

All participants do not use any hormonal contraceptive method.

Exclusion Criteria:

* Participants will be excluded if they had diabetes, hypertension, cardiac diseases, patients who had endocrine disease or digestive tract disease and patients with neurological or musculoskeletal disorder.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Effect of laser acupuncture and abdominal exercises on Body fat mass | 1 cycle (42 days)
  Outcome measurement
Effect of laser acupuncture and abdominal exercises on Body mass index | 1 cycle (42 days)
  Outcome measurement
Effect of laser acupuncture and abdominal exercises on waist girth, hip girth | 1 cycle (42 days)
  Outcome measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Kafar Elsheikh Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No